CLINICAL TRIAL: NCT03381066
Title: A Phase III, Randomized, Multi-center Study to Determine the Efficacy of the Intercalating Combination Treatment of Chemotherapy and Gefitinib or Chemotherapy as Adjuvant Treatment in NSCLC With Common EGFR Mutations.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2016-0763
Record Dates: First submitted 2017-11-22; First posted 2017-12-21 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Completely Resected NSCLC With Common EGFR Mutations
Keywords: NSCLC; EGFR; adjuvant; gefitinib; intercalating
MeSH Terms: interventions — Gefitinib; Pemetrexed; Cisplatin; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intercalating arm (Experimental): gefitinib, pemetrexed,cisplatin
  Interventions: Drug: gefitinib, pemetrexed,cisplatin
- chemotherapy alone arm (Active Comparator): Vinorelbine, cisplatin
  Interventions: Drug: Vinorelbine, cisplatin

INTERVENTIONS:
Drug: gefitinib, pemetrexed,cisplatin — * Intercalation phase (Duration: 3weeks x 4 cycles = 12 weeks) Pemetrexed 500mg/m2 D1, Cisplatin 75mg/m2 D1, Gefitinib 250mg D5-18, every 3week
  * Maintenance phase (Duration: 1 year) Gefitinib 250mg D1-2
  Other Names: Intercalating arm
  Arms: Intercalating arm
Drug: Vinorelbine, cisplatin — Duration: 3wks x 4 cycles = 12 weeks Vinorelbine 25mg/m2 D1,8, Cisplatin 75mg/m2 D1 q3week
  Other Names: chemotherapy alone arm
  Arms: chemotherapy alone arm

SUMMARY:
This study aims to compare the efficacy of intercalating chemotherapy (gefitinib and pemetrexed/cisplatin) and chemotherapy (navelbine/cisplatin) in completely resected NSCLC with common EGFR mutations.

ELIGIBILITY:
Inclusion Criteria:

1. Completely resected non-squamous cell NSCLC with stage IIa to IIIb (excluding N3) according to Version 8 of the IASLC Staging Manual in Thoracic Oncology
2. Tumors with common EGFR mutations (19del or L858R)
3. Adequate oran function

Exclusion Criteria:

1. Patients who were exposed to the chemotherapy or EGFR TKIs for NSCLC.
2. Patients with interstitial lung disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2018-04-10 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
disease-free survival | 5 years
  Time from the randomization to recurrence or any cause of death.

SECONDARY OUTCOMES:
Overall survival | 5 year
  Time from the randomization to death of any cause
Number of participants with treatment-related adverse events as assessed by CTCAE4.0 | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oncology, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided